CLINICAL TRIAL: NCT01591356
Title: EphA2 Gene Targeting Using Neutral Liposomal Small Interfering RNA Delivery: A Phase I Clinical Trial
Brief Title: EphA2 siRNA in Treating Patients With Advanced or Recurrent Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other); Institutional Funding for Federally Supported Clinical Trials (IFSCT) (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0216; NCI-2015-00745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RP120214; NCI-2012-00755; 2011-0216 (Other: M D Anderson Cancer Center); P50CA093459 (NIH)
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (EphA2-targeting DOPC-encapsulated siRNA) (Experimental): Patients receive EphA2-targeting DOPC-encapsulated siRNA IV over 120 minutes on days 1 and 4. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: EphA2-targeting DOPC-encapsulated siRNA; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: EphA2-targeting DOPC-encapsulated siRNA — Given IV
  Other Names: siRNA-EphA2-DOPC
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of EphA2 siRNA in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or have come back after a period of improvement (recurrent). EphA2-targeting DOPC-encapsulated siRNA may slow the growth of tumor cells by shutting down the activity of a gene that causes tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability (toxicity profile) of EphA2-targeting DOPC-encapsulated siRNA (EphA2 siRNA) delivered via neutral liposome (1,2-dioleoyl-sn-glycero-3-phosphatidylcholine or DOPC) administered intravenously in patients with advanced/recurrent malignancies.

II. To determine the maximal tolerated dose (MTD) or maximal administered dose (MAD) using a modified toxicity probability interval (mTPI) design.

SECONDARY OBJECTIVES:

I. To determine efficacy (EphA2 expression modulation) at the MTD or MAD. II. To evaluate the effect of EphA2 siRNA-DOPC on tumor and endothelial cell apoptosis.

III. To record the clinical activity (objective response, duration of response, and time to treatment progression) of intravenous (IV) EphA2 siRNA -DOPC.

IV. To describe the symptom burden of patients receiving siRNA-EphA2-DOPC treatment.

EXPLORATORY OBJECTIVES:

I. To determine the pharmacokinetic profile of siRNA-EphA2-DOPC in blood. II. To determine the effect of EphA2 siRNA-DOPC on tumor perfusion, apparent diffusion, and metabolism by radiographic imaging (dynamic contrast-enhanced-magnetic resonance imaging [DCE-MRI], diffusion weighted [DW]-MRI and fludeoxyglucose F-18-positron emission tomography [18FDG-PET]).

III. To determine the impact of EphA2 siRNA-DOPC on surrogate biomarkers in blood (cell-free deoxyribonucleic acid [DNA], plasma/serum markers [vascular endothelial growth factor (VEGF), caveolin 1 (CAV1), soluble EphrinA1], and exosomes).

OUTLINE: This is a dose-escalation study.

Patients receive EphA2-targeting DOPC-encapsulated siRNA IV over 120 minutes on days 1 and 4. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* All patients with histologic proof of advanced solid tumors, who are not candidates for known regimens or protocol treatments of higher efficacy or priority
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* All patients (dose escalation and dose expansion phases) must be willing to undergo pre- and post-treatment biopsies
* For the dose escalation phase, the trial population will be limited to solid tumor types
* For dose expansion phase: patients must have EphA2 overexpression overall H-score of 3 or above in immunohistochemistry (IHC) evaluation; Clinical Laboratory Improvement Amendments (CLIA) certified EphA2 IHC staining to be performed on formalin fixed, paraffin-embedded tissue sections using monoclonal EphA2 antibody; EphA2 expression to be assessed through a combo of % of positive cells and staining intensity; the % of positive cells will be rated: 0 points (pts), 0 to 5%; 2 pts, 6 to 50%; 3 pts, 50%; the staining intensity will be rated as follows: 1 pt, weak intensity; 2 pts, moderate intensity; 3 pts, strong intensity; pts for expression and % of positive cells will be added; an overall score will be assigned; tumors to be categorized into 4 groups: negative (overall score 0), 5% cells stained, regardless of intensity; weak expression (overall score 1), 1 - 2 pts; moderate expression (overall score 2), 3 - 4 pts; and strong expression (overall score 3), 5 - 6 pts; overall H-score of 3 or above will be defined as EphA2 overexpression in tumor cells
* Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension; at least one biopsiable lesion must be available; when imaging (DCE-MRI, DW-MRI and PET-computed tomography [CT] imaging) is being performed for secondary objectives (dose level III [or when the dose reaches at least 1,500 ug/m^2] and during the expansion phase) at least one lesion (>= 2 cm) not adjacent to the diaphragm will be required when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI; a second lesion accessible for biopsy must also be present; patients must have at least one 'target lesion' to be used to assess response on this protocol as defined by Response Evaluation Criteria in Solid Tumors (RECIST); this may be one of the lesions mentioned above; tumors within a previously irradiated field will be designated as 'non-target' lesions
* Resolution of any effects of prior therapy (except alopecia) to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 grade =< 1 and to baseline laboratory values as defined below
* Hemoglobin (HGB) >= 9 g/dL
* White blood cells (WBC) >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet (PLT) >= 100,000/mcL
* Total bilirubin less than or equal to 1.5
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 2.5 x institutional upper limit of normal (ULN)
* Creatinine < 1.5 x ULN or creatinine clearance > 60 ml/min according to Cockcroft-Gault formula
* Neuropathy (sensory and motor) =< to CTCAE grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is < 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin or low molecular weight heparin) and a partial thromboplastin time (PTT) < 1.2 times control
* Patients should be free of active infection requiring intravenous antibiotics
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration (study enrollment); continuation of hormone replacement therapy is permitted; stable regimens of hormonal therapy i.e. for prostate cancer (e.g. leuprolide, a gonadotropin-releasing hormone [GnRH] agonist), ovarian or breast cancer are not exclusionary
* Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to first dose of study drug (6 weeks for nitrosoureas or mitomycin C)
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for at least 3 months after completion of EphA2 siRNA-DOPC therapy
* Male subject agrees to use an acceptable method of contraception for the duration of the study
* Patients must voluntarily sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital

Exclusion Criteria:

* Patients may not be receiving any other investigational agents and/or other therapy for their cancer
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DOPC, Magnevist, or fluorodeoxyglucose (FDG)
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as a known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases
* Patients with history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study
* Patients with clinically significant cardiovascular disease; this includes: uncontrolled hypertension (greater than 140/90); myocardial infarction or unstable angina within 6 months prior to registration; New York Heart Association (NYHA) grade II or greater congestive heart failure; serious cardiac arrhythmia requiring medication; grade II or greater peripheral vascular disease; patients with clinically significant peripheral artery disease, e.g., those with claudication, within 6 months of first date of treatment on this study
* Patients whose circumstances do not permit completion of the study or the required follow-up
* Patients who are pregnant or nursing
* History of human immunodeficiency virus (HIV) or HIV-positive patients on combination antiretroviral therapy are ineligible
* Patients whose tumor is not accessible for a core biopsy
* Exclusion criteria (MRI specific):

  * Patients who are ineligible to undergo an MRI scan for reasons such as claustrophobia or the presence of implanted devices or metallic foreign bodies that are not magnetic resonance (MR) compatible; patients with a known history of allergic reaction to gadolinium contrast agents; patients with a history of a glomerular filtration rate (GFR) of less than 60 or acute renal disease
* Exclusion criteria (PET specific):

  * Pregnant or nursing women; extreme claustrophobia; weight near or greater than 350 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile of ephrin type-A receptor 2-targeting 1,2-dioleoyl-sn-glycero-3-phosphatidylcholine-encapsulated short-interfering ribonucleic acid | Up to 5 years
  Will be graded according to Common Terminology Criteria for Adverse Events version 4.0
Maximal tolerated dose or maximal administered dose | Up to 21 days
  Will be defined as the dose level with the smallest difference among all tried doses. Will be determined using modified toxicity probability interval design.

SECONDARY OUTCOMES:
Percent of patients with ephrin type-A receptor 2 expression modulation, defined as a 50% decrease from baseline expression | Up to 5 years
  Will be calculated along with 90% exact confidence intervals.
Changes in ephrin type-A receptor 2 expression | Baseline to up to day 4 of course 1
  Tissue effects will be assessed in core biopsy samples collected pre-treatment and course 1 day 2 or day 3 (timed with biomarker assessment).
Changes in endothelial and tumor cell apoptosis conducted by terminal deoxynucleotidyl transferase dUTP nick end labeling assay | Up to 5 years
  Analysis will be performed for both between (dose-effect) and within (changes from baseline) patient cohorts.
Objective response | Up to 5 years
  The best response recorded from the start of the treatment until disease progression/recurrence
Duration of response | Up to 5 years
  measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time to treatment progression | Up to 5 years
  The duration of time from study entry to time of recurrence or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wagner MJ, Mitra R, McArthur MJ, Baze W, Barnhart K, Wu SY, Rodriguez-Aguayo C, Zhang X, Coleman RL, Lopez-Berestein G, Sood AK. Preclinical Mammalian Safety Studies of EPHARNA (DOPC Nanoliposomal EphA2-Targeted siRNA). Mol Cancer Ther. 2017 Jun;16(6):1114-1123. doi: 10.1158/1535-7163.MCT-16-0541. Epub 2017 Mar 6. PMID 28265009
- See also: MD Anderson Cancer Center — http://www.mdanderson.org